CLINICAL TRIAL: NCT07102355
Title: Comparative Effectiveness of Dry Cupping and Graston Techniques in Office Workers With Scapulocostal Syndrome; A Randomised Clinical Trail
Brief Title: Comparative Effectiveness of Dry Cupping and Graston Techniques in Scapulocostal Syndrome.
Acronym: CMR = Compress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Management and Technology Sialkot Pakistan (Other)
Responsible Party: Principal Investigator, Danyal Ahmad, Head Of Department (HOD), University of Management and Technology Sialkot Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: kuhs/dpt/umt-skt-016
Record Dates: First submitted 2024-11-18; First posted 2025-08-03 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Scapulocostal Syndrome
Keywords: Scapulocostal Syndrome; Myofascilal pain syndrome,; Graston Technique; Dry Cupping Therapy; Cervical Range of Motion

STUDY DESIGN:
Intervention Model Description: A convenient sampling technique was used. Data collection was initiated after taking the content form, and then participants were divided into two groups by lottery: Group A and Group B. Group A was given Dry cupping, and Group B was given the Graston Technique along with Conventional Treatment.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A = Dry Cupping (Experimental): Group A will receive Dru cupping along with conventional treatment.
  Interventions: Other: Experimental: Group A = Dry Cupping
- Group B = Graston Technique (Experimental): Group B will receive Graston Technique with Conventional treatment.
  Interventions: Other: Experimental: Group B = Graston Technique

INTERVENTIONS:
Other: Experimental: Group A = Dry Cupping — Dry cupping, originating in Middle Eastern and Asian countries, gained popularity in the United States after the 2016 Summer Olympics. It has two main forms: wet and dry cupping. Wet cupping involves laceration of the skin, while dry cupping uses negative pressure to pull the skin into the cup. Cupping is used to reduce musculoskeletal or myofascial pain, with the most accepted mechanism being localized hyperemia, which improves microcirculation and promotes healing
  Arms: Group A = Dry Cupping
Other: Experimental: Group B = Graston Technique — Instrument-assisted soft tissue mobilization (IASTM), derived from Cyriax cross-friction massage, is a popular alternative to traditional manual therapy techniques, with its first controlled study published in 1997 (Seffrin & Gardiner-Shires, 2019) .The Graston Technique(GT), also known as instrument-assisted soft tissue mobilization (IASTM), is used by chiropractors, doctors, and therapists to alleviate pain and range-of-motion restrictions caused by musculoskeletal injuries and scar tissue. (McKivigan, J. M., & Tulimero, G. et al. , 2020) . The Graston technique, is also used to alleviate upper cervical pain.
  Arms: Group B = Graston Technique

SUMMARY:
The goal of this clinical trial is to check the comparative effectiveness of Graston Techniques and Dry cupping in Office Workers with Scapulocostal syndrome. The main questions it aims to answer are:

1. To evaluate the relative effectiveness of dry cupping and the Graston technique.
2. How well each technique reduces symptoms and enhances work productivity and functional outcomes.
3. To assess whether integrating either Graston Technique or Dry Cupping provides more beneficial effects than conventional treatment alone.

1) Be divided into 2 Groups (Group A= Dry Cupping; B: Graston Techniques) 2) get the treatment for 4 weeks (3 days a week). 3) Receive the same conventional treatment.

DETAILED DESCRIPTION:
This study aims to compare the effectiveness of Graston and Dry cupping in treating Scapulocostal syndrome in office workers, focusing on specific outcomes like pain severity, functional outcomes, and work productivity.

This study will be a randomized clinical trial with a sample size of 46 participants with work-related SCS. The participants will be obtained by non-probability convenient sampling based on the inclusion and exclusion criteria. Participants will be randomly assigned into two groups, with 23 subjects in each group. Group A will receive dry cupping along with conventional therapy while Group B will receive IASTM along with conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18-30 age group
2. Males and females
3. Office Workers.
4. Subjects that have symptoms of musculoskeletal nature (
5. Subjects with pain lasting for longer than 3 months (

Exclusion Criteria:

1. Subjects with underlying pathology such as TOS, brachial neuralgia, cervical radiculopathy, polymyositis or Fibro myositis
2. Subjects with systemic diseases such as rheumatoid arthritis, ankylosing spondylitis
3. Subjects with the presence of any fractures
4. Heart/diabetic patients
5. Pregnant women

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-09-13 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Pain Intensity as Measured by the Visual Analog Scale | 4 Weeks
  Pain intensity will be measured using the Visual Analog Scale (VAS), a 100 mm horizontal line anchored by two extremes: 0 mm represents "no pain" and 100 mm represents "worst imaginable pain." Participants will mark the point that best represents their pain intensity. The score is the distance in millimeters from the left end to the mark. Change in pain intensity will be calculated by subtracting the Week 4 score from the baseline score. A decrease in VAS score indicates an improvement in pain levels.
Cervical Range of Motion (ROM) | 4 weeks
  Cervical spine Range of Motion (ROM) will be assessed and measured using a universal goniometer by utilizing moving and stationary arm of angles in cervical spine range of motion..

SECONDARY OUTCOMES:
Neck Disability Index (NDI) Total Score | 4 Weeks
  The Neck Disability Index (NDI) is a validated 10-item questionnaire assessing neck-specific disability. Each item is scored from 0 to 5, resulting in a total score range of 0 to 50. Higher scores indicate greater disability. The change in total NDI score from baseline to Week 4 will be calculated. A decrease in score indicates clinical improvement.
Treatment-Related Adverse Events During the 4-Week Intervention | 4 weeks
  Treatment-related adverse events (AEs), such as skin irritation, bruising, or discomfort, will be recorded throughout the study. The number of participants experiencing at least one AE will be counted. All AEs will be assessed for severity and relatedness to the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Danyal Ahmad, PhD Scholar, Principal Investigator — University of Management and Technology Sialkot Pakistan
Locations (4):
- Pakistan (4):
  - Bethania Hospital Sialkot, Sialkot, Punjab Province
  - Bethania Hospital, Lahore
  - University of Management and technology Sialkot Campus, Sialkot
  - Bethania Hospital, Sialkot

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) will not be shared, or may not be shared, due to concerns regarding participant confidentiality and privacy, limitations of informed consent that did not explicitly include data sharing, and the risk of re-identification even after anonymization.

REFERENCES:
- [Result] Brandl A, Bartsch K, James H, Miller ME, Schleip R. Influence of Rolfing Structural Integration on Active Range of Motion: A Retrospective Cohort Study. J Clin Med. 2022 Oct 5;11(19):5878. doi: 10.3390/jcm11195878. PMID 36233746
- [Result] Sharma S, Kaur H, Verma N, Adhya B. Looking beyond Piriformis Syndrome: Is It Really the Piriformis? Hip Pelvis. 2023 Mar;35(1):1-5. doi: 10.5371/hp.2023.35.1.1. Epub 2023 Mar 6. PMID 36937215
- [Result] Aslam S, Rahim R, Ejaz U, Tariq ZB, Guftar F. Effects of Myofascial Release Technique on Pain, Range of Motion and Functional Disability in Patients with Piriformis Syndrome. HJPRS [Internet]. 2025 Aug 23 [cited 2025 Oct 19];5(2):56-61.
- [Result] Seffrin CB, Cattano NM, Reed MA, Gardiner-Shires AM. Instrument-Assisted Soft Tissue Mobilization: A Systematic Review and Effect-Size Analysis. J Athl Train. 2019 Jul;54(7):808-821. doi: 10.4085/1062-6050-481-17. Epub 2019 Jul 19. PMID 31322903
- [Result] Buttagat V, Taepa N, Suwannived N, Rattanachan N. Effects of scapular stabilization exercise on pain related parameters in patients with scapulocostal syndrome: A randomized controlled trial. J Bodyw Mov Ther. 2016 Jan;20(1):115-122. doi: 10.1016/j.jbmt.2015.07.036. Epub 2015 Jul 26. PMID 26891646
- [Result] Elsayyad MM, Abdel-Aal NM, Helal ME. Effect of Adding Neural Mobilization Versus Myofascial Release to Stabilization Exercises after Lumbar Spine Fusion: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 Feb;102(2):251-260. doi: 10.1016/j.apmr.2020.07.009. Epub 2020 Aug 19. PMID 32827553